CLINICAL TRIAL: NCT01084200
Title: Comparison of Postoperative Pain of Sevoflurane, Propofol, and Sevoflurane Plus Propofol in Maintenance of Anaesthesia for Gynaecological Laparoscopic Surgery
Brief Title: Comparison of Sevoflurane, Propofol, and Sevoflurane Plus Propofol for Maintenance of Anaesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Wei Mei, Associate Professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TJHMZK01004
Record Dates: First submitted 2010-03-08; First posted 2010-03-10 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Laparoscopic Surgery; Hysteroscopic Surgery
Keywords: Postoperative pain; Sevoflurane; Propofol; Female; Elective gynaecological surgery; Laparoscopic and hysteroscopic surgery; Female patients; Undergoing elective laparoscopic and hysteroscopic surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Propofol; Maintenance; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Propofol (Experimental): anesthesia maintenance with propofol and remifentanil
  Interventions: Drug: Propofol for maintenance
- Sevoflurane (Experimental): Sevoflurane and Remifentanil for anesthesia maintenance
  Interventions: Drug: Sevoflurane
- Sevoflurane+Propofol (Experimental): Sevoflurane+Propofol for anesthesia maintenance
  Interventions: Drug: Sevoflurane+Propofol

INTERVENTIONS:
Drug: Propofol for maintenance — Propofol 6-8mg/kg/h + Remifentail 0.1-0.2ug/kg/min for anesthesia maintenance
  Other Names: Propofol
  Arms: Propofol
Drug: Sevoflurane — Sevoflurane 0.7-1.3MAC + Remifentail 0.1-0.2ug/kg/min for anesthesia maintenance
  Arms: Sevoflurane
Drug: Sevoflurane+Propofol — Sevoflurane 0.7-1.3MAC + Remifentanil 0.1-0.2ug/kg/min + Propofol 2mg/kg/h for anesthesia maintenance
  Other Names: Sevoflurane and Propofol
  Arms: Sevoflurane+Propofol

SUMMARY:
Postoperative pain may be affected by general anaesthetics. The effect of propofol and sevoflurane on postoperative pain in chinese female patients has not been demonstrated before. This study compared the postoperative pain score in patients under general anaesthesia maintained with propofol,sevoflurane, or sevoflurane+propofol.

DETAILED DESCRIPTION:
After approval from the Institute's Ethics Committee, this study was conducted at Tongji Hospital, a general university teaching hospital with 2500 beds in Wuhan, China.The study consisted of female patients, American Society of Anaesthesiologists Physical Status (ASA-PS) I or II, suffering from infertilities, and undergoing selective gynaecological laparoscopic and hysteroscopic surgery. All the patients were randomly assigned to receive propofol,sevoflurane,or sevoflurane+propofol for anaesthesia maintenance. The primary outcome measure was the level of postoperative pain assessed by Numerical Analogue Scale (NAS) at rest 0.5 hour after the operation. The secondary outcomes were postoperative pain assessed by Numerical Analogue Scale (NAS) at rest 1 and 24 hour after the operation, the incidence of postoperative nausea and vomiting, the incidence of shiver, and quality of recovery determined by QOR40 in the first 24 h after surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status class 1 or 2
* Aged >=18 years and =<40 years old
* Suffering from infertilities
* Under elective gynaecological laparoscopic and hysteroscopic surgery

Exclusion Criteria:

* ASA-PS>=III
* Aged under 18 yrs or above 40 yrs old
* Body mass index (BMI) >30
* Respiratory or Neurologic disease
* Chronic antidepressants and Anticonvulsant drugs
* Chronic analgesics intake
* A known allergy to the drugs being used
* History of substance abuse
* Participating in the investigation of another experimental agent
* Participating in the investigation of another study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2009-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Post operative pain determined by NRS at 0.5h after surgery | at 0.5h after the surgery
  The level of postoperative pain was assessed by Numerical Analogue Scale (NAS) at rest at 0.5 hour after the surgery.

SECONDARY OUTCOMES:
Postoperative delirium | 24 hours postoperatively
  Postoperative delirium determined by Nu-DESC every 8 hours.
PONV | 24 hours postoperatively
  Incidence of postoperative nausea and vomiting was assessed at 24h after the surgery.
QOR | 24 hours post operatively
  Quality of recovery was determined by QOR40 at 24h after the surgery
Post operative pain determined by NRS at 1h and 24h after surgery | at 1h and 24h after surgery
  Post operative pain determined by NRS at 1h and 24h after surgery respectively.
Incidence of shivering in the first postoperative day. | follow up at 24 h after the surgery
  Incidence of shivering was assessed at 24h after the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Mei, M.D., Principal Investigator — Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology; Yu Ke Tian, Prof. M.D., Study Chair — Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital, Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Result] Li M, Mei W, Wang P, Yu Y, Qian W, Zhang ZG, Tian YK. Propofol reduces early post-operative pain after gynecological laparoscopy. Acta Anaesthesiol Scand. 2012 Mar;56(3):368-75. doi: 10.1111/j.1399-6576.2011.02603.x. Epub 2011 Dec 23. PMID 22192060